CLINICAL TRIAL: NCT02805881
Title: Safety and Feasibility of Combined Trigeminal and Occipital Transcutaneous Nerve Stimulation (CTO-TNS) in Major Depressive Disorder (MDD)
Acronym: CTO-TNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRLF-BY531-CTIL
Record Dates: First submitted 2016-06-07; First posted 2016-06-20 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurolief System treatment (Experimental): Treatment with the Neurolief system will be applied by the subject at his home and/or surrounding daily during a period of six weeks
  Interventions: Device: Neurolief system

INTERVENTIONS:
Device: Neurolief system — Non-invasive cephalic neurostimulation device

SUMMARY:
Safety and Feasibility of Combined Trigeminal and Occipital Transcutaneous Nerve Stimulation (CTO-TNS) in Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* The subject is capable of understanding the study and to sign an informed consent.
* Subject is between the ages of 18 to 65 years old.
* Unipolar major depressive disorder
* Score on the Hamilton Depression Rating Scale (HDRS21) > 22
* Current MDD episode >3 months
* Nonresponse with >6 week use of one to six antidepressant in current episode

Exclusion Criteria:

* History of neurosurgical interventions.
* Subjects with metal implants or shrapnel in their head, except for dental implants.
* Skin lesion or inflammation at the region of the stimulating electrodes.
* Pregnancy or Lactation.
* Women of reproductive age not using efficient contraceptive method.
* History of cerebrovascular event.
* Psychotic or bipolar depression
* History of schizophrenia, schizoaffective disorder or other non-mood disorder psychosis
* Current delirium, dementia, amnestic disorder or other cognitive disorders
* Clinically significant current suicidal intent as assessed by the investigator team.
* Obsessive-compulsive disorder or post-traumatic stress disorder
* Alcohol and non-alcohol psychoactive substance abuse or dependence
* Significant cardiac, medical, or progressive neurological or medical illness
* An implantable electrical device such as a pacemaker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 weeks
  Safety measures will be recorded and evaluated at every evaluation visit. It will be coded using the Medical Dictionary for Regulatory Activities. Vital signs (blood pressure and pulse) will be assessed and documented at each evaluation visit.
Hamilton Depression Rating Scale (HDRS21) | 6 weeks
  Change in the total score on the Hamilton Depression Rating Scale (HDRS21) from baseline (visit 1) to week 6 (visit 4).

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovitz, Prof., Principal Investigator — Deputy Director, Beer- Yakov Nees-Ziona Mental Health Center
Locations (1):
- Beer- Yakov Nees-Ziona Mental Health Center, Ness Ziona, Israel

IPD SHARING:
Plan to Share IPD: Undecided